CLINICAL TRIAL: NCT02927119
Title: Serum Thyroglobulin as a Marker of Iodine Nutrition Status During Pregnancy in Hungarian Population
Brief Title: Serum Thyroglobulin as a Marker of Iodine Status During Pregnancy
Status: Completed | Type: Observational
Sponsor: University of Debrecen (Other)
Responsible Party: Principal Investigator, Endre V Nagy, Professor, University of Debrecen
Other Study IDs: GRAV-TG
Record Dates: First submitted 2016-10-03; First posted 2016-10-06 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: Dietary Iodine Deficiency; Thyroid; Functional Disturbance
Keywords: thyroglobulin; iodine; pregnancy
MeSH Terms: conditions — Thyroid Diseases | interventions — Iodine

STUDY DESIGN:
Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — serum urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Non-users: Pregnant women who had not taken dietary iodine supplement before and during pregnancy.
- Users: Pregnant women who had taken dietary iodine supplement before and/or during pregnancy.
  Interventions: Dietary Supplement: iodine

INTERVENTIONS:
Dietary Supplement: iodine — ≥ 150 µg/day iodine supplementation (iodine containing pregnancy supplement) prior to enrollment
  Groups: Users

SUMMARY:
The purpose of the investigation is to assess iodine status of pregnant women at week 16 of gestation targeting serum thyroglobulin as a biomarker of iodine deficiency. The investigators aim to assess whether pre-gestational initiation of iodine supplementation is more advantageous in comparison to supplementation start at the time of pregnancy detection.

DETAILED DESCRIPTION:
Mild iodine deficiency is still a public health issue in many industrialized countries, especially during pregnancy. During the last decade there was no monitoring of the iodine status in pregnancy in Hungary.

Since urinary iodine concentration (UIC) only reflects recent iodine intake and carries limited information on individual existing iodine stores, another biomarker e.g. measurement of serum thyroglobulin concentration, would be useful to gain comprehensive information. In the present study, the purpose of the investigation is to compare UIC, UIC normalized to creatinine concentration and serum thyroglobulin as biomarkers of iodine supply in pregnant women in a geographical region where previously iodine deficiency had been found.

UIC, serum thyroglobulin level and thyroid function are measured, and information about iodine supplementation and smoking before and during pregnancy are recorded.

ELIGIBILITY:
Inclusion Criteria:

* healthy pregnant women at week 16 of gestation

Exclusion Criteria:

* thyroid disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women at week 16 of gestation living in Debrecen and its sorroundings
Sampling Method: Probability Sample
Enrollment: 189 (Actual)
Dates: Start 2014-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Urinary iodine concentration | At subject enrollment
  Measurement of urinary iodine concentration (by inductively coupled plasma mass spectrometry) normalized to urine creatinine concentration
Serum thyroglobulin concentration | At subject enrollment
  Measurement of serum thyroglobulin concentration by chemiluminescent immunoassay

SECONDARY OUTCOMES:
Serum thyroid stimulating hormone concentration | At subject enrollment
  Measurement of serum thyroid stimulating hormone concentration by electrochemiluminescence immunoassay
Serum free thyroxine concentration | At subject enrollment
  Measurement of serum free thyroxine concentration by electrochemiluminescence immunoassay
Serum free triiodothyronine concentration | At subject enrollment
  Measurement of serum free triiodothyronine concentration by electrochemiluminescence immunoassay
Serum anti-thyroglobulin autoantibody concentration | At subject enrollment
  Measurement of serum anti-thyroglobulin autoantibody (TgAb) concentration by radioimmunoassay (women with TgAb concentration above 60 IU/L are considered TgAb positive)

CONTACTS AND LOCATIONS:
Overall Officials: Endre V Nagy, MD, PhD, DSc, Principal Investigator — University of Debrecen

IPD SHARING:
Plan to Share IPD: Undecided